CLINICAL TRIAL: NCT01807338
Title: A Follow-up Study on Safety and Tolerability and Pharmacodynamic Effect, of Patients With Idiopathic Parkinson's Disease (PD) of Moderate Severity, Who Have Previously Been Treated With sNN0031, Using an Implanted Catheter and a SynchroMed® II Pump
Brief Title: A Follow-up Study on Safety and Tolerability of Intracerebroventricular Administration of sNN0031 to Patients With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Newron Sweden AB (Industry)
Collaborators: Medtronic (Industry); TFS Trial Form Support (Industry)
Responsible Party: Sponsor
Other Study IDs: sNN0031-002
Record Dates: First submitted 2013-03-07; First posted 2013-03-08 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- saline: Saline administration to patients with idiopathic Parkinson's disease (PD) of moderate severity, who have previously been treated with sNN0031

SUMMARY:
The purpose of this study is to document the long-term safety and tolerability after intracerebroventricular (ICV) administration of sNN0031 (PDGF-BB) in patients who participated in study sNN0031-001

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in study sNN0031-001 with completion of 12 study weeks without development of clinically significant safety concerns, defined as being any drug-related or device related serious adverse event that resulted in premature termination of treatment or a medical device incident that could not be resolved during the conduct of study sNN0031-001
* The patient has a diagnosis of idiopathic PD
* The patient has been given written and verbal information about the follow-up study, has had the opportunity to ask questions about the study, and understands the time and procedural commitments
* The patient has provided written informed consent to participate in the follow-up study

Exclusion Criteria:

* The patient has been included or participates in another clinical study after participation in Study sNN0031-001
* The patient has, since participation in study sNN0031-001, had functional neurosurgical treatment for PD (e.g., deep brain stimulation).
* Patients will only be excluded from participation in the event of a laboratory test abnormality that is indicative of a medical condition requiring treatment which, in the opinion of the investigator, is not compatible with participation in the present study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with idiopathic PD of moderate severity who have completed participation in study sNN0031-001.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2011-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Skåne University Hospital, Lund, Sweden